CLINICAL TRIAL: NCT02894580
Title: Primary Prevention of Sudden Cardiac Death in Real Life: Differences With the Pivotal Studies and Their Consequences
Brief Title: Primary Prevention of Sudden Cardiac Death (PREV-DEATH)
Acronym: PREV-DEATH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-04Obs-CHRMT
Record Dates: First submitted 2016-08-26; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The efficacy of implantable cardioverter-defibrillators (ICD) in primary prevention of sudden cardiac death (SCD) is well demonstrated but pivotal studies have been published more than 10 years ago and implantation's conditions tend to change.

DETAILED DESCRIPTION:
The clinical efficacy of implantable cardioverter defibrillator (ICD) as method of primary prevention of sudden cardiac death (SCD) is well demonstrated today. Unfortunately, selection criteria of patients deemed at risk lacks of specificity. For asymptomatic patients with a left ventricular dysfunction (LVEF), current guidelines support implantation of ICD if the LVEF is ≤35%. This target population corresponds to the one studied in the Sudden Cardiac Death in HEart Failure Trial (SCD-HeFT). This trial is 10 years old. The proportion of patients with LVEF > 30% was low (17%) and the analysis of this subgroup showed no decrease in mortality (hazard ratio = 1.08 [0.57-2.07]). That is why the usefulness of ICD in this segment of the population remains a subject of controversy. Moreover, SCD-HeFT did not offer resynchronization therapy despite the fact that more than 40% of patients included had a QRS signal duration ≥120ms.

Conditions for implantation have since changed considerably. The "routine" nature of the implantation procedure and the desire to maximize patient's protection leads us to address for an implantation more easily. As for the resynchronization, it must be attempted in patients with severe heart failure, LVEF ≤35% and QRS sufficiently prolonged.

This suggests that the implanted population is very different nowadays from those from the pivotal studies in terms of mean LVEF and implanted material. However, these two factors are significantly correlated with the risk of SCD... Therefore, the analysis was done on samples of patients who received ICD in primary prevention setting. This study focused on the effect of resynchronization and LVEF at implantation and the subsequent outcome. The results were broadly compared with those of SCD-HeFT.

ELIGIBILITY:
Inclusion Criteria:

* primo-implantation and primary prevention in New York Heart Association (NYHA) II or III chronic heart failure due to ischemic or non ischemic causes and LVEF ≤35%

Exclusion Criteria:

* Cardiomyopathy other than dilated cardiomyopathy such as hypertrophic cardiomyopathy, congenital or valvular heart disease
* Patients with NYHA class I and IV heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a defibrillator in Metz-Thionville Regional Hospital between January 1, 2009 and December 31, 2014
Sampling Method: Probability Sample
Enrollment: 336 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Mortality from any cause | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michel BOUSIER, MD, Principal Investigator — CHR Metz-Thionville
Locations (1):
- CHR Metz-Thionville, Metz, France

IPD SHARING:
Plan to Share IPD: No